CLINICAL TRIAL: NCT03218111
Title: Evaluation Of Brain Glymphatic Kinetics Following Intrathecal Administration Of Gadolinium In Healthy Adult Volunteers
Brief Title: Glymphatic Kinetics In Healthy Adult Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1609017536
Record Dates: First submitted 2017-07-07; First posted 2017-07-14 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Healthy
Keywords: Glymphatic network; healthy; central nervous system
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy Normal Subjects (Other): Healthy normal subjects 20-80 years old. All subjects will undergo the same procedures: intrathecal injection, using CT-guidance, with an MRI contrast. After injection subjects will undergo six sessions of MR imaging over a 10-12 hour period
  Interventions: Other: MR Imaging; Other: CT-guidance

INTERVENTIONS:
Other: MR Imaging — All subjects will undergo six sessions of MR imaging over a 10-12 hour period
Other: CT-guidance — All subjects will be injected, intrathecally using CT-guidance, with an MRI contrast.

SUMMARY:
This study is being done in order to see how gadolinium-based MRI contrast (Magnevist) travels through the central nervous system (CNS) when injected through the spinal column, and to compare differences between two age groups (age 20-50, and 51-80). This will allow investigators to evaluate how much contrast has crossed into the tissue surrounding the brain. Such information will help investigators determine whether this kind of contrast can be used to model how other drugs might travel through the CNS and evaluate its use as an illustrative imaging marker that mirrors the glymphatic system.

DETAILED DESCRIPTION:
This is a prospective, longitudinal study of MR imaging of intrathecally delivered gadolinium contrast (Magnevist, Gd-DTPA) in healthy adult male and female subjects. Subjects will be divided into two groups (20-50 years old and 51-80 years old) both of which will receive intrathecal injection of the drug Magnevist (Gd-DTPA), followed by serial MR imaging over the course of 10-12 hours. The purpose of the study is determine the transport kinetics of Central Nervous System (CNS) exposure to gadolinium contrast injected into the lumbar intrathecal space (lower back) and evaluate changes with age. This will allow investigators to evaluate the brain parenchymal penetration of gadolinium as an illustrative imaging marker that mirrors the glymphatic system. Investigators hypothesize the exposure and penetration patterns of the neuraxis to neurotherapeutic drugs can be modeled using gadolinium intrathecal contrast administered in the lumbar intrathecal space.

ELIGIBILITY:
Inclusion Criteria:

1. Deemed healthy and able to undergo MR imaging by the Site Investigator, based on screening assessments:

   medical history, physical examination, vital signs, and clinical laboratory values
2. Age 20-80
3. Willing to undergo multiple imaging sessions
4. Normal screening MRI to exclude subjects with a mass (e.g., disk herniation), congenital malformation (e.g., Chiari malformation), or an abnormal curvature of the spine that could alter CSF flow.
5. If female of childbearing age: negative pregnancy test
6. Normal Basic metabolic Panel and CBC (Platelet count > 150,000; Hb >8)
7. Willing to undergo LP procedure. -

Exclusion Criteria:

1. Kyphosis
2. Claustrophobia
3. Chronic cough
4. Active infection with fever (>101.5), to limit risk of meningitis. Infections could include pneumonia, pharyngitis, skin infection, UTI, etc.
5. History of CNS tumor or anomaly
6. History of radiation therapy to the CNS
7. History of hydrocephalus
8. Abnormality on MRI that could impede CSF flow (i.e., extruded disk)
9. Laboratory finding of prolonged coagulation times
10. Pregnant/nursing
11. Prior spine or brain surgery or trauma
12. Inability to lay still and supine
13. Recent lumbar puncture within 1 month of planned LP.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
Drug distribution over time | 6 time-points over 12 hours
  The drug distribution of gadolinium contrast throughout the Central Nervous System over time (12 hours)

CONTACTS AND LOCATIONS:
Overall Officials: J. Levi Chazen, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No Current Plan